CLINICAL TRIAL: NCT06048770
Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of RBI-4000 in Healthy Volunteers
Brief Title: A Study of RBI-4000 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision (not related to safety, efficacy, or quality)
Sponsor: Replicate Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: RBI-4000-101
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Multiple Ascending Dose (MAD) Cohorts, Cohort 1: RBI-4000 0.1 mcg (Experimental): Participants will receive RBI-4000 0.1 micrograms (mcg) via intramuscular injection, once on Day 1 and Day 57.
  Interventions: Biological: RBI-4000
- MAD Cohorts, Cohort 2: RBI-4000 1 mcg (Experimental): Participants will receive RBI-4000 1 mcg via intramuscular injection, once on Day 1 and Day 57.
  Interventions: Biological: RBI-4000
- MAD Cohorts, Cohort 3: RBI-4000 10 mcg (Experimental): Participants will receive RBI-4000 10 mcg via intramuscular injection, single dose on Day 1.
  Interventions: Biological: RBI-4000
- MAD Cohorts, Cohort 4: RBI-4000 10 mcg (Experimental): Participants will receive RBI-4000 ,10 mcg via intramuscular injection, once on Day 1 and Day 57.
  Interventions: Biological: RBI-4000
- Cohort 5: RabAvert 1 mL (Active Comparator): Participants will receive RabAvert 1 milliliter (mL), intramuscular injection, once on Day 1 and Day 8.
  Interventions: Biological: RabAvert

INTERVENTIONS:
Biological: RBI-4000 — RBI-4000 intramuscular injection.
  Arms: MAD Cohorts, Cohort 2: RBI-4000 1 mcg; MAD Cohorts, Cohort 3: RBI-4000 10 mcg; MAD Cohorts, Cohort 4: RBI-4000 10 mcg; Multiple Ascending Dose (MAD) Cohorts, Cohort 1: RBI-4000 0.1 mcg
Biological: RabAvert — RabAvert intramuscular injection.
  Arms: Cohort 5: RabAvert 1 mL

SUMMARY:
The primary purpose of the study is to evaluate the safety, reactogenicity, and immunogenicity of RBI-4000 administered at various dose levels via intramuscular injection and to determine the lowest dose of RBI-4000 necessary to elicit the rabies virus neutralizing antibody titer of equal or greater than (>=) 0.5 international unit per milliliter (IU/mL).

ELIGIBILITY:
Inclusion Criteria:

1. Any gender participants between 18 and 45 years old, inclusive, at the time of the first vaccination.
2. Body Mass Index >18 kilogram per square meter (Kg/m^2) and less than (<) 32 Kg/m^2.
3. Hematological/biochemical values within these parameters:

   1. White Blood Cells and differential, within the study designated laboratory normal range.
   2. Platelets = 125,000 - 500,000 cells per cubic millimeter (cells/mm^3)
   3. Hemoglobin within normal range of the study designated laboratory
   4. Liver function tests including alanine aminotransferase, aspartate aminotransferase, total bilirubin, and alkaline phosphatase within the study designated laboratory normal range.
4. Female participants of non-childbearing potential or male participants with partners of childbearing potential may be enrolled in the study.
5. Female participants of childbearing potential may be enrolled in the study, if the participant

   1. has practiced adequate contraception for 30 days prior to vaccination, and
   2. has a negative pregnancy test on the day of vaccination (for female participants),
   3. has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series and agrees to not donate sperm (for male participants).

Exclusion Criteria:

1. History of diagnosis with rabies exposure, infection or disease.
2. History of rabies immunization (licensed or investigational) or human rabies immune globulin.
3. Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
4. Family history of congenital or hereditary immunodeficiency.
5. History of or current autoimmune disease.
6. History of any reaction or hypersensitivity likely to be exacerbated by any components of commercially available rabies vaccines.
7. Lymphoproliferative disorder or malignancy within previous 5 years (excluding effectively treated non-melanotic skin cancer, Ductal carcinoma in situ /Lobular carcinoma in situ (DCIS/LCIS).
8. History of Type I hypersensitivity reactions to any beta-lactam antibiotics.
9. Any acute or chronic, clinically significant disease, by history, physical examination, laboratory findings, subject personal report, and/or General Physician information.
10. Any history of myocarditis and/or pericarditis.
11. Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
12. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs including steroids during the period within 6 months prior to the vaccine dose.
13. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule.
14. Concomitant or planned administration of antimalarial drugs, including hydroxychloroquine within 30 days of vaccination.
15. Current anti-tuberculosis prophylaxis or therapy.
16. Pregnant or lactating female participant.
17. Female participant planning to become pregnant or planning to discontinue contraceptive precautions.
18. Participants with extensive tattoos covering deltoid region on both the arms that would preclude the assessment of local reactogenicity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of any Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Day 1 up to 18 months
  TEAEs and SAEs measured per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA 2007).
Immunogenicity of RBI-4000 Measured by Neutralizing Antibody Titers | Day 1 up to 18 months
  Measured by neutralizing antibody titers >=0.5 IU/mL.

SECONDARY OUTCOMES:
Titer level of Rabies Virus Neutralizing Antibody | Day 1 and up to 18 months
Durability of RBI-4000 Against Rabies Assessed by T-cell Levels | Day 1 and up to 18 months
  Durability of RBI-4000 against rabies assessed by quantifying cytokine-producing T cells by ELISpot and flow cytometry.
Rate of RBI-4000 Decay Over Time | Day 1 and up to 18 months
Length of Time Above the Recognized Antibody Correlate of Protection Value | Day 1 and up to 18 months
Lowest Dose of RBI-4000 that Provides Durable (greater than [>] 6 months) Coverage Above the Correlate of Protection | Day 1 and up to 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cordova Research Institute, Miami, Florida
  - Velocity Clinical Research, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maine CJ, Picarda G, Miyake-Stoner SJ, Essink B, Somodevilla G, Sparks J, Geall AJ, Wang NS, Goldberg Z, Aliahmad P. Durability of next-generation self-replicating RNA vaccine RBI-4000: a phase 1, randomized open label clinical trial. Commun Med (Lond). 2025 Sep 24;5(1):392. doi: 10.1038/s43856-025-01147-4. PMID 40993199